CLINICAL TRIAL: NCT00913016
Title: Assessment of Quality of Life, Bone Density and Safety in Postmenopausal Breast Cancer Patients With Letrozole (Femara) as an Early Adjuvant Treatment
Brief Title: Assessment of Quality of Life, Bone Density and Safety in Postmenopausal Breast Cancer Patients With Letrozole Therapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Korean Breast Cancer Study Group (Other)
Responsible Party: Sehwan Han, Department of Surgery, Breast Cancer Center, Inje University Paik Hospital
Other Study IDs: KBCSG002
Record Dates: First submitted 2009-05-31; First posted 2009-06-03 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2009-12

CONDITIONS: Breast Cancer
Keywords: hormonal therapy(letrozole); postmenopausal breast cancer; quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- letrozole (Femara)

SUMMARY:
To compare the overall QoL (Quality of Life) using Trial Outcome index (TOI) of FACT-B questionnaire for 3 years from baseline.

DETAILED DESCRIPTION:
1. TOI is the sum of the scores from the physical and functional well-being and the breast cancer subscales.
2. To assess incidence of adverse events (including cardiovascular, cerebrovascular, and endocrine, musculoskeletal) in Korean postmenopausal breast cancer patients in early adjuvant setting.
3. To assess the effect of letrozole (Femara) on BMD in early adjuvant setting.
4. To assess the effect of letrozole (Femara) on total cholesterol in early adjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have undergone surgery of the breast cancer and proven histologically to be breast cancer with postmenopausal women older than 45 years. Postmenopausal state was defined the following conditions, at least one of a, b, c.

   1. serum FSH ≥ 30 mIU/mL
   2. amenorrhea ≥ 1 year
   3. oophorectomy
2. patients with estrogen receptor(+) and/or progesterone receptor(+)
3. WHO(ECOG) performance status 0-2
4. Adequate haematological function, renal function, hepatologic function.
5. No evidence of metastasis.

Exclusion Criteria:

1. patient with hormone receptor negative.
2. Patients with malignancies (other than breast cancer) within the last 5 years, except for adequately treated in situ carcinoma of the cervix or basal cell / squamous cell carcinoma of the skin.
3. Other hormone therapy given within the previous 4 weeks.
4. Patients with other aromatase inhibitor and chemotherapy
5. Uncontrolled infection, medically uncontrollable heart disease
6. Other serious medical illness or prior malignancies
7. Patients with BMD T-score ≤-2.5
8. Patients who were treated with bisphosphonate
9. Patients with postmenopausal state induced chemotherapy
10. Estimated life expectancy of <12 months

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited into the study are postmenopausal women who had undergone surgery for primary breast cancer which was either estrogen receptor(ER) and/or progesteron receptor(PgR)-positive or of both.
Sampling Method: Non-Probability Sample
Enrollment: 897 (Estimated)
Dates: Start 2007-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
overall QoL(Quality of Life) using Trial outcome index(TOI) of FACT-B questionnaire. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sehwan Han, MD.PhD., Principal Investigator — Department of Surgery, Breast Cancer Center,Inje University Paik Hospital, South Korea
Locations (1):
- Department of Surgery, Breast Cancer Center, Inje University Paik Hospital, Seoul, South Korea